CLINICAL TRIAL: NCT03772782
Title: Investigation of the Relationship of Smart Phone Use Addiction With Musculoskeletal System Problems and Cognitive Flexibility
Brief Title: Relationship of SmartPhone Use Addiction With Musculoskeletal System and Cognitive Flexibility
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İNAL, Trakya University, Hacettepe University
Other Study IDs: 09/07
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Smartphone; Musculoskeletal; Cognitive Flexiblity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Smartphones have become a part of everyday life, but with some problems. Researches have pointed out that smartphone addiction can cause both physical and mental problems.

DETAILED DESCRIPTION:
Smartphones have become a part of everyday life, but with some problems. Developments in communication technologies have also improved the capacities and limits of smartphones. This has led to the increased availability of smartphones in daily life. Smartphones have become a part of everyday life, but with some problems. Smartphone addiction has been an important topic of research and discussion as a type of addiction that develops depending on the frequency of smartphone use. Researches have pointed out that smartphone addiction can cause both physical and mental problems. As a result of a study conducted in the literature, continuous use of smartphones has been found to cause sleep disturbances, stress, anxiety, decrease in physical activities and many diseases. In this study, the relationship between the concept of smartphone addiction and musculoskeletal problems and cognitive flexibility in young people will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* University students
* Without any known physical and/or psychological disorders
* Using a smartphone
* Volunteer

Exclusion Criteria:

Have any physical and/or psychological disorders

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: university students between the ages of 18-25
Sampling Method: Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Smartphone addiction scale score | at the end of the third month
  The Smartphone Addiction Scale (SAS) is a33-item, six-point Likert-type self-rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: ÖZGÜ İNAL, Principal Investigator — Trakya University
Locations (1):
- Özgü İnal, Edirne, Turkey (Türkiye)